CLINICAL TRIAL: NCT01530503
Title: A Randomized Phase II Trial of Second Line Therapy in Advanced Biliary Tract Cancer: Capecitabine or Capecitabine Plus Mitomycin C
Brief Title: Second Line Therapy in Advanced Biliary Tract Cancer
Acronym: BIT-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Regione Lombardia (Other)
Responsible Party: Principal Investigator, stefano cereda, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-002002-70
Record Dates: First submitted 2012-02-03; First posted 2012-02-10 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Biliary Tract Cancer
Keywords: biliary tract cancer; advanced disease; chemotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Capecitabine; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- capecitabine (Experimental): oral capecitabine 2000 mg/m2 day 1-14 in two divided doses taken with food
  Interventions: Drug: Capecitabine
- capecitabine plus mitomycin (Experimental): oral capecitabine 2000 mg/m2 day 1-14 in two divided doses taken with food plus bolus IV infusion Mitomycin 6 mg/m2 day 1
  Interventions: Drug: capecitabine and mitomycin

INTERVENTIONS:
Drug: capecitabine and mitomycin — oral capecitabine 2000 mg/m2 day 1-14 in two divided doses taken with food plus bolus IV infusion mitomycin C 6 mg/m2 day 1.
  Cycles will be repeated in both arms every 3 weeks till progression, unacceptable toxicity, medical decision or patient's refusal or for a maximum of 6 months
  Other Names: capecitabine; mitomycin
  Arms: capecitabine plus mitomycin
Drug: Capecitabine — oral capecitabine 2000 mg/m2 day 1-14 in two divided doses taken with food.
  Cycles will be repeated in both arms every 3 weeks till progression, unacceptable toxicity, medical decision or patient's refusal or for a maximum of 6 months
  Arms: capecitabine

SUMMARY:
The purpose of this study is to assess the therapeutic activity of capecitabine alone or in combination with mitomycin C as second-line therapy in patients with advanced/metastatic biliary adenocarcinoma in progression after gemcitabine and platinum compounds

DETAILED DESCRIPTION:
Biliary tract adenocarcinoma is an uncommon tumor with a poor prognosis and a median overall survival (OS) rarely exceeding 6 months. Less than 25% of patients are resectable at diagnosis and, even in this subset of patients, relapse rate is high. An improvement of OS and quality of life for patients receiving chemotherapy versus best supportive care was demonstrated in advanced disease. Recently, cisplatin and gemcitabine combination was identified as the new standard first-line chemotherapy, yielding a median progression free survival (PFS) and median OS of 8.5 and 11.7 months, respectively. Despite the outcome improvement, disease progression is a constant and approximately half of patients failing upfront treatment has a good performance status and are willing to undergo further treatment. No standard salvage chemotherapy regimen has been identified. Clinical trials are difficult to perform due to the rarity and heterogeneity of these tumors and to the lack of interest of the pharmaceutical industry. Fluoropyrimidines and mitomycin C have been considered the basis of palliative chemotherapy for a long time. The investigators decided to explore the activity, in terms of PFS, of capecitabine alone or combined with mitomycin C as second-line therapy in patients with pathological diagnosis of advanced biliary tract cancer and progressive disease after gemcitabine and cisplatin, by means of an open label randomized multicentric phase II trial.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated IRB/IEC-approved Informed Consent.
2. Cytological or histological diagnosis of locally advanced or metastatic adenocarcinoma of the biliary tract (Ampulla of Vater, gallbladder, intra or extra-hepatic biliary ducts).
3. Disease progressing after first-line chemotherapy with gemcitabine and platinum analogs (only one prior systemic therapy allowed).
4. Age 18-75 years
5. Karnofsky Performance Status > 50%
6. Estimated life expectancy of at least 3 months.
7. Negative pregnancy test (if female in reproductive years).
8. Adequate bone marrow, liver and kidney function: leukocyte > 3500/mm3; absolute neutrophil count (ANC) > 1500/mm3; platelet count > 100000/mm3; hemoglobin > 10 g/dl; creatinine < 1.5 mg/dL; total bilirubin ≤ 1.5 x upper limit of normal range (ULN); SGOT e SGPT ≤ 2.5 ULN
9. At the time of start of treatment, at least 2 weeks must have elapsed since completion of prior chemotherapy, minor surgery and radiotherapy (provided that no more than 25% of bone marrow reserve has been irradiated).
10. Resolution of all acute toxic effects of any prior chemotherapy, surgery or radiotherapy to NCI CTC (Version 4.03) grade ≤ 1 for hematologic toxicities and ≤ 2 for non hematologic toxicities, with the exception of alopecia.
11. Able and willing to comply with scheduled visits, therapy plans, and laboratory tests required in this protocol.

Exclusion Criteria:

1. Previous or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-site of the cervix and basal or squamous cell carcinoma of the skin and of other neoplasm without evidence of disease at least from 5 years.
2. Known brain metastases.
3. Previous second-line or adjuvant treatment.
4. Concurrent treatment with other experimental drugs.
5. Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, cardiac arrhythmia) ≤1 year prior to dosing.
6. Clinically significant disease including: Cerebral Vascular Accident; other serious underlying medical condition(s) which could impair the ability of the patient to participate in the study.
7. History of interstitial lung disease (eg, pneumonia or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan
8. Known positive tests for human immunodeficiency virus (HIV) infection, active hepatitis B or hepatitis C
9. Subject who is pregnant or breast feeding
10. Woman or man of child-bearing potential not consenting to use adequate contraceptive precautions ie. double barrier contraceptive methods (e.g., diaphragm plus condom), or abstinence during the course of the study and for 6 months after the last study drug administration for women, and 1 month for men
11. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 6 month PFS
  This is a multi-centre phase II, randomized study. Patients will be stratified based on disease site and stage. For the purpose of the study, PFS-6 rate will be considered the primary outcome measure. The maximum PFS-6 rate of low clinical interest is 15% and the minimum PFS-6 rate of interest is set to 35%. The target enrollment, using a type I error of 5% and a test power of 90%, will be estimated to be 26 patients per treatment arm. The regimen will be considered active if at least 8 out of first 26 evaluable patients are PFS-6.

SECONDARY OUTCOMES:
Overall Survival (OS) | median OS (up to 2 years)
  the time from the date of randomization to the date of death from any cause
  All patients will be followed for survival every 3 months up to 2 years after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: stefano cereda, MD, Principal Investigator — Ospedale San Raffaele (Milan, Italy)
Locations (16):
- Italy (16):
  - ASUR zona territoriale N. 6 FABRIANO, Fabriano, Ancona
  - Fondazione Istituto San Raffaele G. Giglio, Cefalù, Palermo
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I - G.M. Lancisi - G Salesi, Ancona
  - A.O. Ospedali Riuniti, Bergamo
  - Azienda Ospedaliero-Universitaria Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione Piemontese Per la Ricerca sul Cancro, Candiolo (Torino)
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione Garibaldi, Catania
  - Ospedale San Raffaele, Milan
  - Istituto Oncologico Veneto I.R.C.C.S., Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Azienda Ospedaliera Regionale San Carlo, Potenza
  - Istituto Nazionale dei Tumori Regina Elena, Roma
  - Ospedale Generale Provinciale, Saronno (VA)
  - Azienda Ospedaliera Universitaria San Giovanni Battista di Torino, Torino
  - Azienda Ospedaliero Universitaria Santa Maria della Misericordia, Udine
  - Azienda Ospedaliera Universitaria Integrata, Verona